CLINICAL TRIAL: NCT03301636
Title: A Phase 2/3 (Adaptive Design) Study of the Concomitant Administration of Indoximod or Placebo Plus Pembrolizumab or Nivolumab in Adult Patients With Unresectable Stage III or Stage IV Malignant Melanoma
Brief Title: A Study of Indoximod or Placebo Plus Pembrolizumab or Nivolumab for Subjects With Unresectable or Metastatic Melanoma
Acronym: NLG2107
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor termination, not related to efficacy, safety or feasibility.
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NLG2107
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Melanoma
Keywords: Melanoma, Metastaic Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Nivolumab; 1-methyltryptophan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Indoximiod (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Indoximod
- Nivolumab + Indoximiod (Experimental)
  Interventions: Drug: Nivolumab; Drug: Indoximod

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously every 3 weeks starting on day 1.
  Other Names: Keytruda
  Arms: Pembrolizumab + Indoximiod
Drug: Nivolumab — Nivolumab will be administered intravenously every 2 weeks starting on day 1.
  Other Names: Opdivo
  Arms: Nivolumab + Indoximiod
Drug: Indoximod — Indoximod will be administered orally every 12 hours starting at Day 1

SUMMARY:
This is an adaptive clinical trial that includes a dose escalation phase followed by a randomized controlled Phase 3 trial. The purpose of the dose escalation phase is to establish the Phase 3 dose of indoximod in combination with pembrolizumab or nivolumab in subjects with unresectable or metastatic melanoma and evaluate PK. Subsequently the efficacy, safety and tolerability of indoximod plus pembrolizumab or nivolumab versus placebo plus pembrolizumab or nivolumab will be studied in subjects with unresectable or metastatic melanoma in the Phase 3 portion of the trial.

The phase 3 study will not proceed per Sponsor decision.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically- or cytologically-confirmed unresectable stage III or stage IV melanoma not amenable to local therapy
* At least one radiologically measurable lesion as per RECIST 1.1
* Have documentation of V600-activating BRAF mutation status or consent to BRAF V600 mutation testing during the screening period.
* ECOG performance status 0 or 1
* Ability to ingest oral medications

Exclusion Criteria:

* Has Ocular Melanoma
* Has received prior systemic treatment for unresectable or metastatic melanoma (except BRAF directed therapy).
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or IDO1 inhibitor or any other antibody or drug specifically targeting checkpoint pathways other than anti-CTLA-4 which is permitted in the adjuvant setting.
* Has received prior adjuvant therapy, monoclonal antibody or an investigational agent or device within 4 weeks or 5 half-lives (whichever is longer)
* Has received prior radiotherapy within 2 weeks of therapy.
* Is pregnant or breast-feeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.
* Patients who have active, chronic, or on active treatment for Hep B or Hep C are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Utah Cancer Specialists, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Pembrolizumab 200mg Q3 weeks and Indoximod 600mg Q12 hr
- Dose Level 2: Pembrolizumab 200mg Q3 weeks and Indoximod 1200mg Q12 hr
- Dose Level 3: Pembrolizumab 200mg Q3 weeks and Indoximod 1800mg Q12 hr
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 7 | 6 | 8
Completed | 7 | 6 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 7 | 6 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (15.14) | 61.8 (14.77) | 61.9 (8.22) | 61.3 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 12
  Male | 3 | 3 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 6 | 8 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: Centimeters] | 171.3 (10.56) | 168.8 (8.86) | 172.9 (10.25) | 171.1 (9.59)
Weight [Mean (Standard Deviation); unit: Kilograms] | 102.77 (22.3) | 75.12 (13.009) | 117.44 (26.960) | 100.46 (27.502)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Regimen-limiting Toxicities (RLTs) of Indoximod in Combination With Pembrolizumab
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 7 | 6 | 8
Participants | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality (ACM) : Up to ~22.1 months and safety: Up to ~16.5 months
Description: The all-cause mortality and safety were analyzed in all subjects who took at least one dose of study drug. The adverse event table captures treatment-emergent adverse events. In Dose Level 3, 1 of the 8 subjects did not start therapy, resulting in 7 at risk subjects.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 2/7 | 0/6 | 2/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/6 | 3/7
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=7) | Dose Level 2 (N=6) | Dose Level 3 (N=7)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=7) | Dose Level 2 (N=6) | Dose Level 3 (N=7)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 1 (1) | 4 (4)
Pyrexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 6 (6)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Corneal oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT03301636/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT03301636/SAP_001.pdf